CLINICAL TRIAL: NCT00706108
Title: Adaptive Coordination in Anaesthesia Teams and Its Relationship to Clinical Performance. (Cooperative Project ETHZ, OAT, Prof. G. Grote, and IfA/USZ; Founding by Swiss National Science Foundation to Both Institutions)
Brief Title: Adaptive Coordination in Anaesthesia Teams and Its Relationship to Clinical Performance.
Acronym: RACoP
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Johannes Wacker, Institute of Anesthesiology, University Hospital Zurich, University Hospital Zurich
Other Study IDs: SNF 100013-116673 /
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Anesthesia Team Coordination
MeSH Terms: interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Simulation of anesthesia induction with critical incidents: Analysis of technical and non-technical performance (15 Teams)
- 2: Analysis of technical and non-technical performance in live anesthesia inductions (40 teams)
- 3: Simulation of anesthesia inductions with advanced simulated critical incidents or events and analysis of technical and non-technical performance (max. 50 teams)
  Interventions: Behavioral: Observational study

INTERVENTIONS:
Behavioral: Observational study — Observational (descriptive) study of technical and non-technical performance
  Other Names: video analysis
  Groups: 3

SUMMARY:
The impact of different coordination patterns on team performance during anesthesia inductions are analyzed using videotapes. These records are examined using various categorization systems (ETHZ), focussing on changes of coordinative behaviour with shifting situational requirements. A rating system comprising multiple categories is used to evaluate team performance. An integrated simulator study facilitates validation of the rating system.

DETAILED DESCRIPTION:
Video tapes and vital parameter readings are recorded with a setup allowing synchronized recordings. Thus, exact timing between events on different data channels can be determined. Data are analyzed for unforeseen events, technical performance, and team coordination / non-technical performance.

ELIGIBILITY:
Inclusion criteria:

* Anesthesia personnel with at least 3 months practical anesthesia experience
* Patients undergoing surgical procedures

Exclusion criteria:

* Not meeting inclusion criteria
* Lack of consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anesthesia personnel (nurse anesthetists, anesthesia residents, staff anesthetists, OR attendants, other members of anesthesia / perioperative team)and patients as seen on video; all if informed consent was obtained
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2005-01; Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Donat R. Spahn, Prof., MD, Study Director — Institute of Anesthesiology, University Hospital Zurich; Johannes Wacker, MD, Principal Investigator — Institute of Anesthesiology, University Hospital Zurich; Gudela Grote, Prof., PhD, Study Chair — Swiss Federal Institute of Technology ETH Zurich, OAT
Locations (1):
- Institute of Anesthesiology, University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Kunzle B, Zala-Mezo E, Wacker J, Kolbe M, Spahn DR, Grote G. Leadership in anaesthesia teams: the most effective leadership is shared. Qual Saf Health Care. 2010 Dec;19(6):e46. doi: 10.1136/qshc.2008.030262. Epub 2010 May 14. PMID 20472572